CLINICAL TRIAL: NCT06379971
Title: Clinical Trial of Maternal Choline Supplements to Mitigate Effects of Prenatal Cannabis Exposure on Early Brain Development
Brief Title: Maternal Choline Supplementation and Cannabis Use During Pregnancy: Impact on Early Brain Development
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 23-2327
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Child Development; Cannabis Use
Keywords: phosphatidylcholine; choline
MeSH Terms: interventions — Rice Bran Oil; Choline; Phosphatidylcholines

STUDY DESIGN:
Intervention Model Description: Phosphatidylcholine versus placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will take 8 placebo capsules each containing 1100mg Rice Bran Oil and 150mg Pumpkin Seed Oil every day in place of phosphatidylcholine supplement.
  Interventions: Drug: Placebo
- Phosphatidylcholine (Active Comparator): Participants will take 8 900mg capsules of phosphatidylcholine every day, the equivalent of approximately 1028 mg of choline per day until delivery
  Interventions: Drug: Choline

INTERVENTIONS:
Drug: Placebo — Pregnant women are instructed to take the capsules twice per day, 4 placebo capsules at breakfast and 4 placebo capsules at dinner. Increased awareness of the benefits of choline by obstetricians and pregnant women, as well as our published results from an observational study showing a wide distribution of plasma choline concentration, is a more apt independent variable for analyses.
  Other Names: rice bran oil and pumpkin seed oil
  Arms: Placebo
Drug: Choline — Pregnant women are instructed to take the capsules twice per day, 4 900mg phosphatidylcholine capsules at breakfast and 4 capsules at dinner. Increased awareness Increased awareness of the benefits of choline by obstetricians and pregnant women, as well as our published results from an observational study showing a wide distribution of plasma choline concentration, is a more apt independent variable for analyses.
  Other Names: Phosphatidylcholine
  Arms: Phosphatidylcholine

SUMMARY:
The goal of this study is to determine if providing a nutritional supplement, phosphatidylcholine, to pregnant women who have used cannabis products during the current pregnancy improves the offspring's brain-related development during the first 3 months. Participating pregnant women will receive either phosphatidylcholine or a placebo from approximately 16 weeks gestation through birth. The primary outcomes are the child's brain responses to sound at 4 weeks corrected age and infant behaviors at 3 months corrected age as reported by the primary caregiver. Secondary outcomes include motor, socio-emotional, language and cognitive development.

DETAILED DESCRIPTION:
Phosphatidylcholine (PC) is a form of choline, a nutrient that is sometimes referred to as Vitamin B4 or Vitamin J. Choline is for normal growth everywhere in the body, including in the brain. PC is a naturally occurring substance and can be found in many different kinds of food including milk, liver, and eggs so most people get enough choline. However, when a woman is pregnant and her baby is growing many new cells, more PC may be needed. Research has suggested that the presence of adequate amounts of choline during pregnancy and breastfeeding can help ensure healthy fetal brain development and may have long-lasting positive effects on cognitive function. Problems in behavioral and cognitive development into childhood have been reported in children of mothers who used cannabis during gestation. Alternatively, two studies of maternal choline levels during pregnancy have reported beneficial effects of higher levels on childhood behavioral and cognitive development. This study assesses whether a higher dose of choline taken during pregnancy will have positive results on offspring development.

Participants in this double-blind study will be randomly assigned to receive either placebo or 1028 mg of choline daily throughout pregnancy, until delivery. Vital signs will be taken, potential side effects will be assessed, and study medication will be given at each visit. Blood samples will be taken at enrollment, and approximately at weeks 16, 22, 28, 34. Children will be followed and assessed until 3 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who report cannabis use during current pregnancy

Exclusion Criteria:

* Pregnancies complicated by fetal anomaly, including neural tube defect or chromosomal abnormality, or multiple gestations due to increased obstetrical risks
* Women with major preexisting maternal medical morbidities
* Women with a prior history of fetal death
* Current personal history of chronic infections, including HIV
* Current personal or family history out to first-degree relatives of trimethylaminuria or homocystinuria
* Primary language other than English or Spanish
* Evidence of noncompliance

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Infant Behavior Questionnaire-Revised (IBQ-R) Orienting/Regulation Index | 3 months corrected age
  The Orienting/Regulation Index is derived by adding the maternal rating of the infant's duration of attention, distractibility, soothability, cuddling, and smiling on the 91-item IBQ-r
Auditory Sensory Gating (P50) | 1 month corrected age
  Inhibition of the P50 cerebral auditory evoked response is collected during a paired stimulus auditory sensory gating paradigm

SECONDARY OUTCOMES:
Maternal Plasma Choline Levels | approximately 16, 22, 28, 34 weeks gestation
  Plasma choline levels will be used to assess the effects of supplementation throughout gestation
Bayley Scales of Infant and Toddler Development | 1, 3 and 6 months corrected age
  The Bayley Scales are a standardized assessment of language, cognitive and motor development
Child Behavior Checklist (CBCL) 1 1/2-5 | 18 months corrected age
  The CBCL assesses a wide range of parent reported behaviors in children on a normative scale for comparison with others, including those assessed in need of clinical interventions for behavioral problems

CONTACTS AND LOCATIONS:
Overall Officials: M. Camille Hoffman, MD, Principal Investigator — University of Colorado, Denver; Sharon Hunter, PhD, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- UC Health, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes